CLINICAL TRIAL: NCT03827889
Title: Efficacy of Two Protocols for Applying Fluorine Varnish to Initial Active Lesions of Deciduous Teeth: a Randomized Clinical Trial
Brief Title: Efficacy of Two Protocols for Applying Fluorine Varnish to Deciduous Teeth
Acronym: CEPECO3
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Outbreak of COVID-19.
Sponsor: Universidade Ibirapuera (Other)
Responsible Party: Principal Investigator, Tamara Kerber Tedesco, PhD, Senior Lecturer, Universidade Ibirapuera
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIB5
Record Dates: First submitted 2019-01-22; First posted 2019-02-04 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Dental Caries
Keywords: dental caries; Tooth, Deciduous; Fluorides, Topical
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WMP of fluoride varnish (Experimental): Whole mouth protocol group
  Interventions: Procedure: WMP of fluoride varnish
- TWLP of fluoride varnish (Experimental): Tooth with lesion Protocol
  Interventions: Procedure: TWLP of fluoride varnish
- DHP (educational intervention) (Active Comparator): Diet and Hygiene guidance Protocol
  Interventions: Behavioral: DHP (educational intervention)

INTERVENTIONS:
Procedure: WMP of fluoride varnish — Application of fluoride varnish (drug of the intervention - Duraphat, Colgate) on all teeth, regardless of the lesions found
  Arms: WMP of fluoride varnish
Procedure: TWLP of fluoride varnish — application of the fluoride varnish (drug of the intervention - Duraphat, Colgate) only on the teeth with active initial caries lesions detected through visual examination after prophylaxis
  Arms: TWLP of fluoride varnish
Behavioral: DHP (educational intervention) — The control group will receive diet and hygiene guidance (educational intervention) through verbal explanations and teeth brushing practices
  Arms: DHP (educational intervention)

SUMMARY:
Evidence that the data flow analysis tests, there are still no studies that show the clarity of the protocols of its application, including the interval and execution factors of applications, concentration of fluoridation and previous prophylaxis. That is, there are still large gaps regarding fluoride varnish applications. Thus, the objective of the present project is the selection of two protocols for application of fluid applications in active drugs in primary tooth enamel. The longitudinal follow-up will be performed in a period of 3, 6, 12, 18 and 24 months after the procedure. The progression of a subject will be evaluated clinically through the transition of ICDAS scores and assessment of the lesions (sound examination with superficial measurements) by visual examination, and the physician evaluates the efficacy and the ability to evaluate the therapeutic techniques and evaluation. treatment, cost and quality of life of participants

ELIGIBILITY:
Inclusion Criteria:

* Children with active carious lesions scores 1, 2 or 3 of the ICDAS in deciduous teeth

Exclusion Criteria:

* Patients with special needs;
* Patients using orthodontic appliances;
* systemic diseases;
* Teeth that present restorations, sealants, formation defects, deep caries lesions that may lead to pulp involvement, fistulae and / or abscesses;
* teeth with spontaneous painful symptomatology.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
PROGRESSION OF CARIES LESIONS (caries lesions inactivation assessment) | Every 6 months up to 24 months
  Caries progression will be evaluated radiographically by three previously trained evaluators (through theoretical classes and evaluation of 13 clinical photographs) and calibrated. These examiners will not know the chronological order and compare the images two to two first by two evaluators and when there is disagreement between the two, the third examiner shall be called for tie-breaker. The possible progression of the treated caries lesion will be codified as:
  * Present progression: Change in radiolucidity area of the Lesion
  * Absent progression: No change in the area of radiolucidity of the lesion.

SECONDARY OUTCOMES:
Number of surfaces with NEW CARIES LESIONS | Up to 24 months
  Detection of the presence of new lesions in deciduous and permanent teeth through visual inspection after dental cleaning. New lesions will be recorded using ICDAS scores.
Children self-reported discomfort | baseline (Immediately after procedure)
  The child's discomfort will be assessed immediately after the sequence of treatments performed in each session by the Wong-Baker face scale. Each face corresponds to a number in a numeric scale from 0 to 5, being 0 no discomfort and 5 maximum of discomfort. At the end, the averages of each score will be compared between the experimental groups.The patient will be asked to choose the face that is more similar to how he/she felt during the treatment. The answer should be given solely by the child, which means no parental or professional interferences.
COST-EFFICACY of each protocol | up to 24 months
  To evaluate the cost-efficacy of different protocols by total value in dollar of treatment in relation to efficacy.The quantities of all consumables used in each procedure will be annotated, as well as the time spent in each procedure, money and time will be combined to report the cost of procedures, measured by $/hour. In addition, we will verify the efficacy through the need for new surgical treatments or new caries lesions. In this way, we will compare the experimental groups according to the cost ($/hour) x the efficacy (need for new interventions). The costs of each treatment procedure will be calculated and compared with thresholds values for intervention by region, determined by World Health Organization (http://www.who.int/choice/costs/CER_levels/ en/).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Ibirapuera, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available on Mendeley database